CLINICAL TRIAL: NCT05114642
Title: Evaluation of the Effect of Face Mask Treatment on Head Posture, Pharyngeal Airway, Skeletal and Dental Structures in Patients With Maxillary Retrognathia
Brief Title: The Effect of Orthopedic Face Mask Use on Head Posture and Pharyngeal Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taner OZTURK, DDS, MS (Other)
Responsible Party: Sponsor-Investigator, Taner OZTURK, DDS, MS, Lecturer, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/669
Record Dates: First submitted 2021-10-19; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Class III Malocclusion; Hyoid Bone
Keywords: Class III Malocclusion; Craniocervical Posture; Hyoid Bone Position; Pharyngeal Airway
MeSH Terms: conditions — Malocclusion, Angle Class III | interventions — Palatal Expansion Technique

STUDY DESIGN:
Intervention Model Description: Head posture on lateral cephalometric radiographs taken before and after the application of the rapid maxillary expansion device with hooks to the upper dental arch and the Petit type face mask treatment applied after the skeletal class III patients due to maxillary retrognathia, whose growth development continues, for treatment to the Orthodontics Department of the Faculty of Dentistry, cervical posture, pharyngeal airway, and hyoid bone positions are determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skeletal Class III Malocclusion Treatment with Face Mask Group (Experimental): In patients with skeletal class III malocclusion (ANB angle < 0,0) due to maxillary deficiency, rapid maxillary expansion appliances prepared on dental plaster models made of acrylic material covering all the upper dental posterior tooth surfaces were applied before the upper jaw was orthopedically brought forward with a face mask. This process was stopped when the expansion was made so that the palatal tubercles of the maxillary permanent first molars align with the buccal tubercles of the mandibular permanent first molars. Immediately afterwards, the petit-type face mask was applied to the hooks of the maxillary expansion device with the help of elastic bands and used continuously for at least 18 hours a day. After obtaining a positive overjet, the face mask appliance was used at night to ensure retention, and then the treatment was terminated.
  Interventions: Device: Skeletal Class III Malocclusion Treatment with Face Mask Group
- Control Group (No Intervention): A control group was formed from patients in the same age group who had skeletal class III malocclusion due to maxillary growth deficiency but were not treated. In this way, the changes that occurred in the normal process in the head, craniocervical postures, pharyngeal airway and hyoid bones of the patients whose growth and development continued could be distinguished.

INTERVENTIONS:
Device: Skeletal Class III Malocclusion Treatment with Face Mask Group — Expanding the maxilla, which is narrower than the mandible in the transverse dimension, using a rapid maxillary expansion device and protraction of the maxilla, which is located behind in the sagittal dimension, forward using the face-mask appliance.
  Other Names: Maxillary expansion
  Arms: Skeletal Class III Malocclusion Treatment with Face Mask Group

SUMMARY:
The aim of this study was to evaluate the changes in head posture, position of the hyoid bone, pharyngeal airway and cervical posture after the use of Petit type face mask in patients with skeletal class III malocclusion (ANB angle < 0) with ongoing growth.

No other study was found in the literature in which head posture, cervical posture, and hyoid bone position were evaluated after the use of a face mask and compared with a control group consisting of patients of the same age group and the same malocclusion.

DETAILED DESCRIPTION:
All radiographic assessments, including cephalometric, pharyngeal airway and craniocervical measurements were performed by the same researcher and she was blind to all the treatment details, orthodontic records, and information of the subjects to prevent bias. Lateral cephalometric radiographs were taken digitally with an X-ray unit (OP300; Instrumentarium Dental, Tuusula, Finland) according to the manufacturer and same technician. Subjects were positioned at the natural head position, teeth in centric occlusion, and lightly closed lips for lateral cephalometric radiographs. Skeletal development of individuals was evaluated using cervical vertebra maturation method (Ref: Bacetti T., An Improved Version of the Cervical Vertebral Maturation (CVM) Method for the Assessment of Mandibular Growth. Angle Orthod.). The skeletal development of individuals was evaluated using the cervical vertebra maturation method and it was determined that all patients were in the prepubertal stage (CS1-CS3). (Ref: Cevidanes L., Comparison of two protocols for maxillary protraction: bone anchors versus face mask with rapid maxillary expansion. Angle Orthod.)

ELIGIBILITY:
Inclusion Criteria:

* For the study group it is as follows:

  1. Patients with skeletal Class III association (ANB < 0°)
  2. Maxillary insufficiency patients
  3. Patients with ongoing growth development
  4. Patients who have used a 'Petit type face mask' for anterior positioning of the maxilla
* For the control group it is as follows:

  1. Patients with skeletal Class III association (ANB < 0°)
  2. Maxillary insufficiency patients
  3. Patients with ongoing growth development
  4. Patients who have not had any orthodontic treatment

Exclusion Criteria:

1. Patients with a congenital anomaly or a craniofacial deformity
2. Patients who have undergone orthodontic treatment
3. Patients with tooth extraction or tooth loss
4. Patients with a history of trauma
5. Patients who have completed growth development (patients with Ru on wrist film)

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Craniocervical posture change | Before treatment (T0) and after treatment (up to about 10-12 month; T1) for the study group. First measurement (T0) for the control group and after similar follow-up time (up to about 10-12 month; T1) as for the treatment group.
  Investigation of the change in head posture after treatment of class III malocclusion due to maxillary deficiency with a face mask using craniocervical angles (NSL/CVT, NSL/OPT, CVT/HOR, OPT/HOR, NL/VER, NSL/VER).
Pharyngeal airway change | Before treatment (T0) and after treatment (up to about 10-12 month; T1) for the study group. First measurement (T0) for the control group and after similar follow-up time (up to about 10-12 month; T1) as for the treatment group.
  Investigation of the change in pharyngeal airway dimensions after treatment of class III malocclusion due to maxillary deficiency with a face mask using pharyngeal airway sagittal dimension measurements (PNS-UPW, Cv2-MPW, Cv3-LPW, HRL/U-PNS, U-PNS, PASmin).
Hyoid bone position change | Before treatment (T0) and after treatment (up to about 10-12 month; T1) for the study group. First measurement (T0) for the control group and after similar follow-up time (up to about 10-12 month; T1) as for the treatment group.
  Investigation of the change in hyoid bone position after treatment of class III malocclusion due to maxillary deficiency with a face mask using hyoid bone location measurements (H-Cv2, H-Cv3, H-Mandibular line, H-Me).

SECONDARY OUTCOMES:
Correlation of craniocervical posture, pharyngeal airway and hyoid bone change | Before treatment (T0) and after treatment (up to about 10-12 month; T1) for the study group. First measurement (T0) for the control group and after similar follow-up time (up to about 10-12 month; T1) as for the treatment group.
  Investigation of the relationship between changes in craniocervical posture, pharyngeal airway dimensions and hyoid bone position.

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Coban, DDS, MDS, Principal Investigator — Erciyes University, Faculty of Dentistry, Department of Orthodontics
Locations (1):
- Erciyes University Faculty of Dentistry, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solow B, Sandham A. Cranio-cervical posture: a factor in the development and function of the dentofacial structures. Eur J Orthod. 2002 Oct;24(5):447-56. doi: 10.1093/ejo/24.5.447. PMID 12407940
- [Background] Gul Amuk N, Kurt G, Baysal A, Turker G. Changes in pharyngeal airway dimensions following incremental and maximum bite advancement during Herbst-rapid palatal expander appliance therapy in late adolescent and young adult patients: a randomized non-controlled prospective clinical study. Eur J Orthod. 2019 May 24;41(3):322-330. doi: 10.1093/ejo/cjz011. PMID 30892615
- [Background] Kilinc AS, Arslan SG, Kama JD, Ozer T, Dari O. Effects on the sagittal pharyngeal dimensions of protraction and rapid palatal expansion in Class III malocclusion subjects. Eur J Orthod. 2008 Feb;30(1):61-6. doi: 10.1093/ejo/cjm076. Epub 2007 Sep 28. PMID 17906307